CLINICAL TRIAL: NCT07217613
Title: Prospective Evaluation of Silk Fibroin Incision Dressings in ACL Reconstruction: A Biocompatible Alternative for High-Motion Surgical Sites
Brief Title: Prospective Evaluation of Silk Fibroin Incision Dressings in ACL Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25-01002
Record Dates: First submitted 2025-10-15; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Silk fibroin adhesive incision dressing (Experimental): Participants will receive the silk fibroin adhesive incision dressing following anterior cruciate ligament reconstruction (ACLR).
  Interventions: Device: silk fibroin-based incision dressing
- Standard closure dressing (Active Comparator): Participants will receive the standard-of-care incision management currently used in ACL reconstruction at NYU Langone Orthopedic Surgery, consisting of cyanoacrylate-based closure systems (e.g., Dermabond® or Prineo®) as determined by the operating surgeon.
  Interventions: Device: cyanoacrylate-based closure system
- Bilateral procedures (Experimental): For bilateral procedures (contralateral patellar tendon harvest for autograft), a within-subject design will be employed: one incision site will receive silk fibroin and the other cyanoacrylate, with side assignment randomized.
  Interventions: Device: silk fibroin-based incision dressing; Device: cyanoacrylate-based closure system

INTERVENTIONS:
Device: silk fibroin-based incision dressing — Applied sterile, hydrophobic, hypoallergenic dressing remains in place for 14-21 days, unless removal is clinically indicated (e.g., saturation, detachment, suspected allergic contact dermatitis, or at provider discretion).
  Other Names: SYLKE®; SYLKE Inc.
  Arms: Bilateral procedures; Silk fibroin adhesive incision dressing
Device: cyanoacrylate-based closure system — Applied per standard NYU practice; dressing remains in place per routine protocol.
  Other Names: Dermabond®; Prineo®
  Arms: Bilateral procedures; Standard closure dressing

SUMMARY:
The purpose of this study is to compare the incidence of early postoperative skin complications including allergic contact dermatitis, blistering, and erythema between silk fibroin incision dressings and cyanoacrylate mesh closure in patients undergoing anterior cruciate ligament reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 to 60 years
* Scheduled for primary or revision ACL reconstruction (ACLR)
* Able and willing to provide informed consent (≥18 years) or assent with parental/guardian permission (ages 14-17)
* Able and willing to comply with all study-related procedures and follow-up visits

Exclusion Criteria:

* Active dermatologic conditions at or near the surgical site (e.g., eczema, psoriasis, dermatitis, open wounds)
* Immunocompromised state (e.g., uncontrolled HIV, ongoing chemotherapy, chronic corticosteroid therapy)
* Known or suspected allergy or hypersensitivity to silk fibroin or cyanoacrylate adhesives
* Uncontrolled diabetes (defined as most recent HbA1c ≥ 8.0, if available; not measured for study purposes)
* Active tobacco use within 30 days of surgery
* Active systemic infection at the time of enrollment

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-10-14 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of postoperative skin complications (allergic contact dermatitis, blistering, erythema) | Follow-up 1 (7-14 days postoperatively)

SECONDARY OUTCOMES:
Percentage of participants with intact dressing | Follow-up 2 (4-6 weeks postoperatively)
Participant reported comfort rating as assessed by the Visual Analogue Scale (VAS) | Follow-up 2 (4-6 weeks postoperatively)
  Patients will complete a 0-10 VAS rating for comfort.
Participant reported itch rating as assessed by the VAS | Follow-up 2 (4-6 weeks postoperatively)
  Patients will complete a 0-10 VAS rating for itch.
Rehabilitation Interference score | Follow-up 2 (4-6 weeks postoperatively)
  A 5-point Likert scale (none → extreme) will assess the perceived impact of incision-related discomfort on physical therapy participation and return to activity.
Overall participant satisfaction rating as assessed by the VAS | Follow-up 2 (4-6 weeks postoperatively)
  Patients will complete a 0-10 VAS rating for comfort.
Participant perceived scar quality score as assessed by the Patient and Observer Scar Assessment Scale (POSAS) | ~4-6 months postoperative
  POSAS v2.0 is validated for evaluating scar quality, including pigmentation, pliability, thickness, and overall cosmetic outcome. The scale consists of 6 items rated from 1 to 10. The total score ranges from 6 to 60. A score of 6 represents normal skin, while a score of 60 indicates the worst imaginable scar. The overall opinion question is rated separately and is not included in the total score.
Participant perceived scar quality score as assessed by the Patient and Observer Scar Assessment Scale (POSAS) | ~1 year postoperative
  POSAS v2.0 is validated for evaluating scar quality, including pigmentation, pliability, thickness, and overall cosmetic outcome. The scale consists of 6 items rated from 1 to 10. The total score ranges from 6 to 60. A score of 6 represents normal skin, while a score of 60 indicates the worst imaginable scar. The overall opinion question is rated separately and is not included in the total score.
Number of dressing-related complications requiring intervention | Day 30
  Assessed via electronic medical record (EMR) review.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a single-site, minimal-risk device study. Only aggregate results will be disseminated; individual datasets will not be shared. The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: layne.estes@nyulangone.org or ivanka.bhambani@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.